CLINICAL TRIAL: NCT07344779
Title: ROAD - Real-World Outcomes of Darolutamide, ADT, With or Without Docetaxel in Metastatic Hormone-Sensitive Prostate Cancer
Brief Title: A Study to Learn How Men With Advanced Prostate Cancer Respond to Treatment With Darolutamide and Hormone Therapy, With or Without Chemotherapy, in Real-world Medical Practice
Acronym: ROAD
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23100
Record Dates: First submitted 2025-12-15; First posted 2026-01-15 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Hormone-Sensitive Prostate Cancer
Keywords: Prostatic Neoplasms, Hormone-Sensitive/Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide; Docetaxel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Darolutamide + ADT + Docetaxel (Triplet therapy): This group includes men with metastatic hormone-sensitive prostate cancer (mHSPC) who are treated with a combination of darolutamide, androgen deprivation therapy (ADT), and docetaxel. The decision to use this triplet therapy is made by the treating physician as part of routine clinical practice before the patient enrolls in the study. Patients in this cohort receive all three treatments according to local standard of care.
  Interventions: Drug: Darolutamide (BAY 1841788); Drug: ADT; Drug: Docetaxel
- Darolutamide + ADT (Doublet therapy): This group includes men with metastatic hormone-sensitive prostate cancer (mHSPC) who are treated with darolutamide and androgen deprivation therapy (ADT), but without docetaxel. The decision to use this doublet therapy is made by the treating physician as part of routine clinical practice before the patient enrolls in the study. Patients in this cohort receive darolutamide and ADT according to local standard of care.
  Interventions: Drug: Darolutamide (BAY 1841788); Drug: ADT

INTERVENTIONS:
Drug: Darolutamide (BAY 1841788) — Darolutamide administered per local standard of care in combination with ADT.
  Other Names: NUBEQA
Drug: ADT — Androgen deprivation therapy administered per local standard of care.
Drug: Docetaxel — Docetaxel administered per local standard of care in combination with darolutamide and ADT for cohort 1.
  Groups: Darolutamide + ADT + Docetaxel (Triplet therapy)

SUMMARY:
This is an international, prospective, open-label, multicenter, multi-cohort, non-interventional observational study designed to describe the real-world effectiveness and safety of darolutamide in combination with androgen deprivation therapy (ADT), with or without docetaxel, in patients with metastatic hormone-sensitive prostate cancer (mHSPC). The study aims to enroll approximately 1,600 male patients (800 per cohort) from multiple countries, primarily in Europe, who have a diagnosis of mHSPC and for whom a decision to treat with darolutamide has been made by the treating physician prior to enrollment. The primary objective is to estimate the proportion of patients achieving undetectable prostate-specific antigen (PSA) levels (<0.2 ng/mL) at 1 year of treatment in each cohort. Secondary objectives include describing patient demographics, clinical characteristics, prior and concomitant treatments, adverse events, and clinical effectiveness measures such as overall survival, time to new treatment, time to castration resistance, and time to PSA progression. Further objectives involve assessing quality of life, reasons for not adding docetaxel, outcomes by patient subgroups (e.g., Gleason score, disease volume, ECOG status), genomic testing results, and hospitalization rates. Data will be collected using electronic case report forms (eCRF) during routine clinical practice, with no additional diagnostic or monitoring procedures required beyond standard care. All patients must provide informed consent prior to participation. The study will comply with applicable regulatory requirements, including IEC/IRB approval in all participating countries. Statistical analyses will be descriptive and exploratory, with interim analyses planned after 200, 400, and 600 patients per cohort have completed at least 12 months of treatment or discontinued therapy. The study is expected to provide valuable insights into the real-world use of darolutamide in mHSPC, supporting clinical decision-making and enhancing understanding of treatment patterns, effectiveness, and safety in diverse patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Male patient with a diagnosis of mHSPC
* Male aged ≥18 years (or country's legal age of adulthood if >18 years)
* Histologically or cytologically confirmed adenocarcinoma of prostate; may have begun ADT (up to 120 days prior to enrollment)
* Metastatic disease by conventional or new generation imaging
* Decision to initiate treatment with darolutamide with or without docetaxel made prior to enrollment
* Signed informed patient consent before start of data collection
* Life expectancy of ≥3 months based on clinical judgment

Exclusion Criteria:

* Participation in an investigational program with interventions outside of routine clinical practice
* Contraindications according to local marketing authorization
* Any prior treatment with second-generation AR inhibitors (enzalutamide, apalutamide, or investigational AR inhibitors), CYP17 inhibitors (abiraterone acetate or investigational CYP17 inhibitors) as antineoplastic treatment for prostate cancer
* Prior hormone therapy in the metastatic setting
* Treatment with darolutamide initiated more than 7 days prior to enrollment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with a diagnosis of metastatic hormone-sensitive prostate cancer (mHSPC) for whom a decision to treat with darolutamide has been made by the treating physician prior to enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in cohort 1 achieving undetectable PSA (<0.2 ng/mL) at 1 year | after 1 year of treatment
  To describe the effectiveness of darolutamide + ADT + docetaxel in patients with mHSPC by means of estimating the prostate-specific antigen (PSA) undetectable rates (PSA<0.2 ng/mL) after 1 year of study treatment.
Proportion of patients in cohort 2 achieving undetectable PSA (<0.2 ng/mL) at 1 year | after 1 year of treatment
  To describe the effectiveness of darolutamide + ADT in patients with mHSPC by means of estimating the prostate-specific antigen (PSA) undetectable rates (PSA<0.2 ng/mL) after 1 year of study treatment.

SECONDARY OUTCOMES:
Overall survival per cohort and per country | up to 4 years
  Time from start of darolutamide treatment until death from any cause.
Overall survival per cohort in all countries | up to 4 years
  Time from start of darolutamide treatment until death from any cause.
Time to subsequent treatment per cohort and per country | up to 4 years
  Time from start of darolutamide treatment to initiation of a new anti-cancer therapy.
Time to subsequent treatment per cohort in all countries | up to 4 years
  Time from start of darolutamide treatment to initiation of a new anti-cancer therapy.
Time to castration resistance (CRPC) per cohort and per country | up to 4 years
  Time from enrollment until documented clinical or PSA progression with testosterone level <50 ng/dL or documented medical/surgical castration.
Time to castration resistance (CRPC) per cohort in all countries | up to 4 years
  Time from enrollment until documented clinical or PSA progression with testosterone level <50 ng/dL or documented medical/surgical castration.
Time to PSA progression per cohort and per country | up to 4 years
  Time from start of darolutamide treatment to PSA progression (≥25% increase above nadir and ≥2 ng/mL, confirmed by a second value ≥3 weeks later, but prior to 6 months, while on treatment).
Time to PSA progression per cohort in all countries | up to 4 years
  Time from start of darolutamide treatment to PSA progression (≥25% increase above nadir and ≥2 ng/mL, confirmed by a second value ≥3 weeks later, but prior to 6 months, while on treatment).
PSA response rate per cohort and per country | 1 year
  Proportion of patients with blood PSA level <0.2 ng/mL, confirmed by a second subsequent PSA value <0.2 ng/mL 3 or more weeks later
PSA response rate per cohort in all countries | 1 year
  Proportion of patients with blood PSA level <0.2 ng/mL, confirmed by a second subsequent PSA value <0.2 ng/mL 3 or more weeks later
Survival rate per cohort and per country | up to 4 years
  Survival rate at specified time points.
Survival rate per cohort and all countries | up to 4 years
  Survival rate at specified time points.
Time to discontinuation per cohort and per country | up to 4 years
  Time from start of darolutamide treatment to permanent discontinuation or death
Time to discontinuation per cohort in all countries | up to 4 years
  Time from start of darolutamide treatment to permanent discontinuation or death
Reason for discontinuation percohort and per country | up to 4 years
  Reason for permanent darolutamide discontinuation
Reason for discontinuation per cohort in all countries | up to 4 years
  Reason for permanent darolutamide discontinuation
Patient demographics per cohort and per country | at baseline
  Demographic characteristics at the first documented regular visit ion the study, referred to as baseline).
Patient demographics per cohort in all countries | at baseline
  Demographic characteristics at the first documented regular visit ion the study, referred to as baseline).
Medical History per cohort and per country | at baseline
  The medical history will be documented at study start.
Medical History per cohort in all countries | at baseline
  The medical history will be documented at study start.
Concomitant medication per cohort and per country | up to 4 years
  Documentation of Concomitant medication.
Concomitant medication per cohort in all countries | up to 4 years
  Documentation of Concomitant medication.
Concomitant treatment per cohort and per country | up to 4 years
  Documentation of Concomitant treatments.
Concomitant treatment per cohort in all countries | up to 4 years
  Documentation of Concomitant treatments.
Darolutamide use per cohort and per country | up to 4 years
  To describe real-world use of darolutamide in mHSPC patients.
Darolutamide use per cohort in all countries | up to 4 years
  To describe real-world use of darolutamide in mHSPC patients.
Diagnostic Imaging Technology per cohort and per country | at baseline
  Documentation of Diagnostic Imaging Technology at the initial study visits (baseline).
Diagnostic Imaging Technology per cohort in all countries | at baseline
  Documentation of Diagnostic Imaging Technology at the initial study visits (baseline).
Adverse events per cohort and per country | up to 4 years
  Number of all adverse events.
Adverse events per cohort in all countries | up to 4 years
  Number of all adverse events.
Serious Adverse events per cohort and per country | up to 4 years
  Number of all serious adverse events.
Serious Adverse events per cohort in all countries | up to 4 years
  Number of all serious adverse events.
Drug-related Adverse events per cohort and per country | up to 4 years
  Number of all drug-related (darolutamide) adverse events.
Drug-related Adverse events per cohort in all countries | up to 4 years
  Number of all drug-related (darolutamide) adverse events.
Serious Drug-related Adverse events per cohort and per country | up to 4 years
  Number of all serious drug-related (darolutamide) adverse events.
Serious Drug-related Adverse events per cohort in all countries | up to 4 years
  Number of all serious drug-related (darolutamide) adverse events.
Adverse events leading to treatment discontinuation per cohort and per country | up to 4 years
  Number of adverse events leading to treatment discontinuation.
Adverse events leading to treatment discontinuation per cohort in all countries | up to 4 years
  Number of adverse events leading to treatment discontinuation.
Vital Signs: Blood Pressure per cohort and per country | up to 4 years
  Blood Pressure is measured in mmHg throughout the study, at all major visit types, over the full observation period.
Vital Signs: Blood Pressure per cohort in all countries | up to 4 years
  Blood Pressure is measured in mmHg throughout the study, at all major visit types, over the full observation period.
Vital Signs: Body Temperature per cohort and per country | up to 4 years
  Body Temperature is measured in degrees Celsius (°C) or Fahrenheit (°F) (as per local practice) throughout the study, at all major visit types, over the full observation period.
Vital Signs: Body Temperature per cohort in all countries | up to 4 years
  Body Temperature is measured in degrees Celsius (°C) or Fahrenheit (°F) (as per local practice) throughout the study, at all major visit types, over the full observation period.
Vital Signs: Weight per cohort and per country | up to 4 years
  Weight is measured in kilograms (kg) throughout the study, at all major visit types, over the full observation period.
Vital Signs: Weight per cohort in all countries | up to 4 years
  Weight is measured in kilograms (kg) throughout the study, at all major visit types, over the full observation period.
Vital Signs: Height per cohort and per country | up to 4 years
  Height is measured in centimeters (cm) throughout the study, at all major visit types, over the full observation period.
Vital Signs: Height per cohort in all countries | up to 4 years
  Height is measured in centimeters (cm) throughout the study, at all major visit types, over the full observation period.
Laboratory Parameters: Hematology (Hemoglobin) per cohort and per country | up to 4 years
  Hemoglobin (g/dL)) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Hematology (Hemoglobin) per cohort in all countries | up to 4 years
  Hemoglobin (g/dL)) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Hematology (WBC) per cohort and per country | up to 4 years
  White Blood Cell Count (WBC) (x10^9/L) is performed throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Hematology (WBC) per cohort in all countries | up to 4 years
  White Blood Cell Count (WBC) (x10^9/L) is performed throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Hematology (Platelet Count) per cohort and per country | up to 4 years
  Platelet Count (x10^9/L) is performed throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Hematology (Platelet Count) per cohort in all countries | up to 4 years
  Platelet Count (x10^9/L) is performed throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (Creatinine) per cohort and per country | up to 4 years
  Serum Creatinine (mg/dL or µmol/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (Creatinine) per cohort in all countries | up to 4 years
  Serum Creatinine (mg/dL or µmol/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (ALT) per cohort and per country | up to 4 years
  Alanine Aminotransferase (ALT) (U/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (ALT) per cohort in all countries | up to 4 years
  Alanine Aminotransferase (ALT) (U/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (AST) per cohort and per country | up to 4 years
  Aspartate Aminotransferase (AST) (U/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (AST) per cohort in all countries | up to 4 years
  Aspartate Aminotransferase (AST) (U/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (Bilirubin) per cohort and per country | up to 4 years
  Total Bilirubin (mg/dL or µmol/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (Bilirubin) per cohort in all countries | up to 4 years
  Total Bilirubin (mg/dL or µmol/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (Alkaline Phosphatase) per cohort and per country | up to 4 years
  Alkaline Phosphatase (U/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (Alkaline Phosphatase) per cohort in all countries | up to 4 years
  Alkaline Phosphatase (U/L) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (PSA) per cohort and per country | up to 4 years
  Prostate-Specific Antigen (PSA) (ng/mL) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.
Laboratory Parameters: Clinical Chemistry (PSA) per cohort in all countries | up to 4 years
  Prostate-Specific Antigen (PSA) (ng/mL) is determined throughout the study, at all major visit types, for the duration of darolutamide treatment and as needed during follow-up, up to the end of observation.

CONTACTS AND LOCATIONS:
Locations (16):
- Many Locations, Multiple Locations, Belgium
- Many Locations, Multiple Locations, Finland
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Greece
- Many Locations, Multiple Locations, Israel
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Lithuania
- Many Locations, Multiple Locations, Norway
- Many Locations, Multiple Locations, Poland
- Many Locations, Multiple Locations, Portugal
- Many Locations, Multiple Locations, Saudi Arabia
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Sweden
- Many Locations, Multiple Locations, Switzerland
- Many Locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Currently, there is no established plan for the sharing of Individual Patient Data (IPD) from this study. The availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA 'Principles for responsible clinical trial data sharing.' This pertains to the scope, timepoint, and process of data access. As such, Bayer commits to considering requests from qualified researchers for patient- / study-level clinical trial data, and documents from clinical trials involving medicines and indications approved in the US and EU. However, this commitment does not reflect an active IPD sharing plan. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Researchers can use www.vivli.org to request access to IPD and documents from clinical studies to conduct research. Information on Bayer's criteria for listing studies is provided in the member section of the portal.